CLINICAL TRIAL: NCT03474198
Title: Two-month Regimens Using Novel Combinations to Augment Treatment Effectiveness for Drug-sensitive Tuberculosis
Acronym: TRUNCATE-TB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National University Hospital, Singapore (Other); Singapore Clinical Research Institute (SCRI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRUNCATE-TB
Record Dates: First submitted 2018-03-12; First posted 2018-03-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin; Isoniazid; Pyrazinamide; Ethambutol; Linezolid; Clofazimine; rifapentine; Levofloxacin; bedaquiline

STUDY DESIGN:
Intervention Model Description: This study uses a multi-arm, multi-stage (MAMS) parallel study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard TB Management Strategy (Active Comparator): Standard combination treatment for pulmonary TB of 8 weeks rifampicin, isoniazid, pyrazinamide, ethambutol, then 16 weeks rifampicin, isoniazid only
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol
- TRUNCATE-TB Management Strategy using Regimen B (Experimental): TRUNCATE-TB Management Strategy: 8 weeks* of initial treatment using Regimen B; close monitoring after treatment completion; treatment of relapse with 24 weeks of standard treatment.
  *If persistent symptoms and positive smear at week 8, extend to 12 weeks of treatment using Regimen B; if persistent symptoms and positive smear at week 12, switch to standard treatment regimen and extend to 24 weeks of treatment.
  Regimen B: Rifampicin (35mg/kg), isoniazid, pyrazinamide, ethambutol, linezolid
  Interventions: Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Linezolid; Drug: Rifampicin
- TRUNCATE-TB Management Strategy using Regimen C (Experimental): TRUNCATE-TB Management Strategy as described above, using Regimen C in place of B.
  Regimen C: Rifampicin (35mg/kg), isoniazid, pyrazinamide, ethambutol, clofazimine
  Interventions: Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Clofazimine; Drug: Rifampicin
- TRUNCATE-TB Management Strategy using Regimen D (Experimental): TRUNCATE-TB Management Strategy as described above, using Regimen D in place of B.
  Regimen D: Rifapentine, isoniazid, pyrazinamide, linezolid, levofloxacin
  Interventions: Drug: Isoniazid; Drug: Pyrazinamide; Drug: Linezolid; Drug: Rifapentine; Drug: Levofloxacin
- TRUNCATE-TB Management Strategy using Regimen E (Experimental): TRUNCATE-TB Management Strategy as described above, using Regimen E in place of B.
  Regimen E: Isoniazid, pyrazinamide, ethambutol, linezolid, bedaquiline
  Interventions: Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Drug: Linezolid; Drug: Bedaquiline

INTERVENTIONS:
Drug: Rifampicin — 10mg/kg
  Arms: Standard TB Management Strategy
Drug: Isoniazid — 5mg/kg
Drug: Pyrazinamide — 25mg/kg
Drug: Ethambutol — 15mg/kg
  Arms: Standard TB Management Strategy; TRUNCATE-TB Management Strategy using Regimen B; TRUNCATE-TB Management Strategy using Regimen C; TRUNCATE-TB Management Strategy using Regimen E
Drug: Linezolid — 600mg
  Arms: TRUNCATE-TB Management Strategy using Regimen B; TRUNCATE-TB Management Strategy using Regimen D; TRUNCATE-TB Management Strategy using Regimen E
Drug: Clofazimine — 200mg
  Arms: TRUNCATE-TB Management Strategy using Regimen C
Drug: Rifapentine — 1200mg
  Arms: TRUNCATE-TB Management Strategy using Regimen D
Drug: Levofloxacin — 1000mg
  Arms: TRUNCATE-TB Management Strategy using Regimen D
Drug: Bedaquiline — 400mg once daily for 2 weeks then 200mg 3x a week
  Arms: TRUNCATE-TB Management Strategy using Regimen E
Drug: Rifampicin — 35mg/kg
  Arms: TRUNCATE-TB Management Strategy using Regimen B; TRUNCATE-TB Management Strategy using Regimen C

SUMMARY:
The current standard management strategy for drug-sensitive pulmonary tuberculosis (TB) is to treat with multiple drugs for 6 months, although patients often fail to adhere to the long treatment, leading to poor clinical outcomes including drug resistance, which is expensive and difficult to treat.

The TRUNCATE-TB trial evaluates an alternative strategy (the TRUNCATE-TB Management Strategy) comprising treatment for 2 months (8 weeks, extended to 12 weeks if inadequate clinical response) with a regimen predicted to have enhanced sterilising activity ("boosted regimen") and monitoring closely after treatment cessation. Those who relapse (predicted to be always drug sensitive and likely to occur early) will be retreated with a standard 6 month regimen.

The trial is a randomized, open-label, multi-arm, multi-stage (MAMS) trial to test the hypothesis that the TRUNCATE-TB Management Strategy is non-inferior to the standard management strategy in terms of longer-term outcomes (clinical status at 96 weeks). If non-inferiority is demonstrated then the advantages/disadvantages of implementing the strategy will be explored in secondary outcomes (from patient and programme perspective).

The trial will evaluate the TRUNCATE-TB Management Strategy with 4 potential boosted regimens (180 per arm, total 900 with the standard TB management strategy arm). The boosted regimens include new drugs (licensed drugs, repurposed from other indications) and optimized doses of standard drugs, selected based on consideration of maximal sterilising effect, absence of drug-drug interactions, as well as safety and tolerability over a period of 2 months

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Clinical symptoms consistent with pulmonary TB and/or evidence of pulmonary TB on chest X-ray (CXR)
3. Sputum GeneXpert test positive
4. Willing to comply with the study visits and procedures
5. Resident at a fixed address
6. Willing to have directly observed therapy
7. Willing and able to provide written informed consent

Exclusion Criteria:

1. Taken more than 10 daily doses of standard anti-TB medication or fluoroquinolones during the 3 months prior to randomisation
2. Previous active TB disease for which treatment was given prior to the current episode
3. Known or suspected extra-pulmonary TB
4. Severe clinical pulmonary TB
5. Sputum smear 3+ on microscopy*
6. Cavity size > 4cm on screening CXR*
7. Presence of rifampicin resistance on GeneXpert test
8. Poorly-controlled diabetes that, in the opinion of the investigator, is unlikely to be controlled with available management strategies
9. Active malignancy requiring systemic chemotherapy or radiotherapy
10. Known Hepatitis B surface antigen positive and/or HCV antibody positive, unless liver function tests consistently within normal range for at least 2 years
11. History of myocardial infarction, congestive cardiac failure, cardiac arrhythmias or any known congenital cardiac problems
12. History of severe chronic lung disease with symptom score of ≥3 on MRC breathlessness scale
13. History of seizures
14. Current tendinitis or history of tendinopathy associated with fluoroquinolone use
15. Symptomatic peripheral neuropathy causing greater than minimal interference with usual social and functional activities
16. Current alcohol or drug abuse
17. Women who are currently pregnant or breast-feeding
18. Women of childbearing potential unwilling or unable to use appropriate effective contraception for the first 6 months of the trial
19. Known allergy to one or more of the study drugs
20. Taking a concomitant medication that has a known or predicted interaction with any of the study drugs to which the patient might be randomised, or is known to prolong the QTc interval
21. Taking any immunosuppressive drugs or use of systemic corticosteroids for more than 2 weeks prior to screening
22. Colour blindness detected by Ishihara test

23.12-lead ECG at screening shows QTc greater than 450ms and/or any other clinically-significant abnormality such as arrhythmia or ischaemia

24.Any of the following laboratory parameters at screening:

* Absolute neutrophil <1000 cells/mL, haemoglobin <7.0 g/dL, OR platelet count <50,000 cells/mm3
* Creatinine clearance of <60ml/min (calculated using Cockcroft-Gault equation)
* ALT greater than 3 times the upper limit of normal
* Uncorrected serum potassium <3.5 mmol/L

  25.HIV antibody positive at screening*

  26.Any other significant condition (e.g. psychiatric illness, chronic diarrhoeal disease), that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial or lead to poor compliance with study visits and protocol requirements

  27.Participation in other clinical intervention trial or research protocol

Note: *Criteria may be modified in later stages of the trial

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Unsatisfactory clinical outcome at week 96 after randomisation | 96 weeks
  As defined by ongoing requirement for TB treatment at week 96 OR ongoing TB disease activity at week 96 (clinical, microbiological and/or imaging evidence) OR death before week 96

SECONDARY OUTCOMES:
Acceptability of the strategy using trial-specific questionnaire | 96 weeks
  7-item trial-specific questionnaire
Total days on TB drug treatment | 96 weeks
Time off work or study due to illness/treatment | 96 weeks
Total Quality of life using MOS-HIV questionnaire | 96 weeks
  MOS-HIV questionnaire
Respiratory disability at week 96 | 96 weeks
Total Grade 3 or 4 clinical adverse events | 96 weeks
Total serious adverse events | 96 weeks
Death | 96 weeks
Adherence to TB medication | Either during first 8 weeks or at any time during period when TB treatment is prescribed
Treatment default | Either during first 8 weeks or at any time during period when TB treatment is prescribed
Acquired drug resistance by week 96 | 96 weeks
Community transmission risk | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Study Director — National University Hospital, Singapore
Locations (18):
- National Institute of TB and Respiratory Diseases, New Delhi, India
- Indonesia (5):
  - Universitas Padjadjaran, Bandung
  - Persahbahatan Hospital, Jakarta
  - Wahidin Sudirohusodo Hospital, Makassar
  - Saiful Anwar Hospital, Malang
  - Soetomo General Hospital, Surabaya
- Philippines (6):
  - Perpetual Succour Hospital, Cebu
  - De La Salle Health Sciences Institute, Manila
  - Lung Center Philippines, Manila
  - Philippines Tuberculosis Society Incorporated (PTSI), Manila
  - Tropical Disease Foundation, Manila
  - Quezon Institute, Quezon City
- National University Hospital, Singapore, Singapore
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Central Chest Institute of Thailand, Nonthaburi
- Uganda (3):
  - Infectious Diseases Institute, Kampala
  - Joint Clinical Research Centre, Kampala
  - Joint Clinical Research Centre, Mbarara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paton NI, Cousins C, Sari IP, Burhan E, Ng NK, Dalay VB, Suresh C, Kusmiati T, Chew KL, Balanag VM, Lu Q, Ruslami R, Djaharuddin I, Sugiri JJR, Veto RS, Sekaggya-Wiltshire C, Avihingsanon A, Saini JK, Papineni P, Nunn AJ, Crook AM; TRUNCATE-TB Trial Team. Efficacy and safety of 8-week regimens for the treatment of rifampicin-susceptible pulmonary tuberculosis (TRUNCATE-TB): a prespecified exploratory analysis of a multi-arm, multi-stage, open-label, randomised controlled trial. Lancet Infect Dis. 2025 Oct;25(10):1084-1096. doi: 10.1016/S1473-3099(25)00151-3. Epub 2025 May 22. PMID 40414233
- [Derived] Paton NI, Cousins C, Suresh C, Burhan E, Chew KL, Dalay VB, Lu Q, Kusmiati T, Balanag VM, Lee SL, Ruslami R, Pokharkar Y, Djaharuddin I, Sugiri JJR, Veto RS, Sekaggya-Wiltshire C, Avihingsanon A, Sarin R, Papineni P, Nunn AJ, Crook AM; TRUNCATE-TB Trial Team. Treatment Strategy for Rifampin-Susceptible Tuberculosis. N Engl J Med. 2023 Mar 9;388(10):873-887. doi: 10.1056/NEJMoa2212537. Epub 2023 Feb 20. PMID 36808186
- [Derived] Converse PJ, Almeida DV, Tasneen R, Saini V, Tyagi S, Ammerman NC, Li SY, Anders NM, Rudek MA, Grosset JH, Nuermberger EL. Shorter-course treatment for Mycobacterium ulcerans disease with high-dose rifamycins and clofazimine in a mouse model of Buruli ulcer. PLoS Negl Trop Dis. 2018 Aug 13;12(8):e0006728. doi: 10.1371/journal.pntd.0006728. eCollection 2018 Aug. PMID 30102705